CLINICAL TRIAL: NCT04358705
Title: C-FLASH (Cigarillo Flavor and Abuse Liability, Attention, and Substitution in youtH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CASE13Z19
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Smoking Behaviors
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Young Cigarillo User (YCU) Sample (Experimental): Aim 1: Online survey. 392 participants from the full YCU sample
  Supplemental Aim 1: A sample of 196 heterosexual females from the Aim 1 survey will be compared to the SGM females
  Aim 2: 150 participants from Columbus, Ohio, and surrounding areas will be recruited for an Eye Tracking Activity to capture visual attention to cigarillo packaging. Visual attention will be examined in 3 conditions: 1) flavored product images, 2) unflavored product images, and 3) a mixture of flavored and unflavored product images.
  Aim 3: (162 participants from Aim 1 survey). Consists of the Online Electronic Tobacco Marketplace (ETM) and the aim 3 survey components:
  * Demographic screener questions
  * Tobacco product withdrawal scale
  * ETM
  * Quality Assurance Question
  * Tobacco product withdrawal scale
  * Survey (nicotine dependence & flavor preferences)
  A sample of 88 from the 162 Aim 3 participants will be compared with 88 SGM participants from supplemental Aim 1.
  Interventions: Other: Aim 1: Online survey; Behavioral: Eye Tracking Activity; Other: Eye tracking survey; Behavioral: Online Experimental Marketplace (ETM); Other: Aim 3 survey; Other: Supplemental Aim 1 Interviews
- Sexual and Gender Minority (SGM) Female Cigarillo Users (Experimental): Supplemental Aim 1: An online convenience sample of 196 SGM females will complete the Aim 1 online survey and will be compared to sample of 196 heterosexual females from the YCU sample
  Supplemental Aim 3: (88 SGM females who participated in the Supplemental Aim 1 survey). Consists of the ETM and the aim 3 survey components in the following order:
  * Demographic screener questions
  * Tobacco product withdrawal scale
  * ETM
  * Quality Assurance Question
  * Tobacco product withdrawal scale
  * Survey (nicotine dependence & flavor preferences)
  Interventions: Other: Aim 1: Online survey; Behavioral: Eye Tracking Activity; Other: Eye tracking survey; Behavioral: Online Experimental Marketplace (ETM); Other: Aim 3 survey
- Cognitive interview (Other): Separate population of participants (n=29) who were a mix of cigarillo users, dual e-cigarette and cigarillo users, e-cigarette users, and non-users. The cognitive interviews informed the Aim 1 survey
  Interventions: Other: Cognitive Interviews

INTERVENTIONS:
Other: Aim 1: Online survey — This survey will evaluate perceptions of flavors on appeal, purchasing and risk perceptions of cigarillo products among young adult and adolescent cigarillo users. This survey will be used to inform survey design for further aims.
  As a proxy for biological verification of tobacco use status, data on brand, frequency, and pricing will be collected to confirm user status
  Participants will rate the role of flavor and report perceptions of product appeal, health risk, advertising exposure and use intentions. Participants will also complete purchase and substitution tasks.
  Arms: Sexual and Gender Minority (SGM) Female Cigarillo Users; Young Cigarillo User (YCU) Sample
Behavioral: Eye Tracking Activity — The eye tracking activity consists of a single in-person eye tracking activity that will take place in a private office in Columbus, Ohio where the participant will be seated in a chair within a typical viewing distance from a computer monitor equipped with an infrared camera on the monitor to capture precise eye movements. Participants will have their gaze monitored continuously by the camera on the computer monitor while a randomized set of stimuli (e.g., tobacco product images) are viewed (n=30) for 10 seconds per image. Following each image, an on-screen closed response question will re-center the participant's gaze for standardization prior to the next image.
  Arms: Sexual and Gender Minority (SGM) Female Cigarillo Users; Young Cigarillo User (YCU) Sample
Other: Eye tracking survey — Other Names: Participants will complete a survey using Qualtrics immediately after the eye tracking activity and one week following completion of the activity via email to measure recall of brand name, product flavors, perceptions of cigarillo harm, and tobacco use behaviors and intentions.
  Arms: Sexual and Gender Minority (SGM) Female Cigarillo Users; Young Cigarillo User (YCU) Sample
Behavioral: Online Experimental Marketplace (ETM) — Administered online via Qualtrics
  Participants are given an account balance for use during their assigned ETM based on their average weekly tobacco use calculated from previous interview. Participants will view all four price conditions and all four flavor conditions in random order for a total of 16 rounds
  Cigarillo price conditions: 1) market price 2) ½ market price 3) 2X market price 4) 4X market price
  Flavor condition: 1) flavored cigarillos and fruit-flavored disposable-cigarettes available 2) unflavored cigarillos and fruit-flavored ecigarettes available 3) flavored cigarillos and tobacco-flavored e-cigarettes available 4) unflavored cigarillos and tobacco-flavored e-cigarettes available.
  Participants will purchase cigarillos with their account balance. During all ETM conditions, constant-priced alternative tobacco products (smokeless tobacco, nicotine lozenges, nicotine gum, and the nicotine patch) will be available in addition to the cigarillos and e-cigarettes.
  Arms: Sexual and Gender Minority (SGM) Female Cigarillo Users; Young Cigarillo User (YCU) Sample
Other: Aim 3 survey — Consists of:
  * A screener and demographic data collection.
  * A tobacco product withdrawal scale
  * Upon completion of the ETM, participants will be asked to respond to a quality assurance question regarding the conditions that varied. Participants will be shown a list of 8 possible conditions and must chose one of the three that varied in order to be eligible to receive compensation.
  * The tobacco product withdrawal scale again
  * Measurements of nicotine dependence and flavor preferences
  Arms: Sexual and Gender Minority (SGM) Female Cigarillo Users; Young Cigarillo User (YCU) Sample
Other: Cognitive Interviews — Cognitive Interviews will be done in-person, using Zoom, or over the phone. Interviews will be video or audio recorded. . The participant will be given a select section of the survey questions from Aim 1. The survey will be uploaded to Qualtrics to reflect the way that survey would be conducted in Aim 1. With the survey questions in front of the participant on the computer screen, research personnel will ask probing questions about each one of the survey questions. If the participant is not able to participate in person or via Zoom, they will be allowed to be interview over the phone with access to the Qualtrics survey or a paper form. If the participant is unable to access the internet, the participant will be read the questions by research personnel. The participant will provide feedback about the questions and walk the research personnel through their thought process for approaching each survey question.
  Arms: Cognitive interview
Other: Supplemental Aim 1 Interviews — Participants from the preceding online survey (who identify as women from Aim 1/supplemental aim 1 survey) who agreed to be contacted for future study will be emailed an invitation to the eligibility screener. Individuals interested will complete a screener to ensure participants identify as women and to verify that they have ever used cigarillos. Eligible participants will be contacted to schedule a 60- to 90-minute Zoom interview about their tobacco, nicotine, and cannabis product use experiences, with particular focus on flavored cigarillo usage initiation, current use, and responses to potential flavor restrictions.
  Arms: Young Cigarillo User (YCU) Sample

SUMMARY:
The purpose of this research is to understand how flavor affects young adult's perceptions of little cigar or cigarillo use.

DETAILED DESCRIPTION:
The overall goal of this study is to examine and better understand adolescent and young adult perceptions, visual attention, use intentions and purchasing behaviors among users and non-users of cigarillos.

Supplemental Aim 1: Consists of evaluation of the differences in perceptions of flavors on appeal, purchasing and risk perceptions of cigarillo products between young adult sexual and gender minorities (SGM) and heterosexual females. A convenience sample of SGM females will be recruited using online social media platforms with targeted advertising. From the parent survey (or Aim 1), an existing sample of female heterosexual cigarillo users will be leveraged. Both samples will receive the same survey, Aim 1, to compare perceptions of appeal, risk, and purchasing across cigarillos and other tobacco products.

Aim 1 of this study is exploratory and will consist of an online survey. Findings from Aim 1 will inform the questions asked about advertising and product use in Aim 2 and 3. Both Aim 2 and 3 are randomized sections. Participants in Aim 2 are either tobacco users or non-users. Participants will be asked to view a series of tobacco related images. The sequence of those images is randomized. In Aim 3, participants will be randomized in terms of the options they are presented within the Experimental Tobacco Marketplace (ETM) (i.e. which tobacco items they can purchase and at what price).

Supplemental Aim 3 consists of evaluating the differences in the abuse liability/addictive potential of flavored versus unflavored cigarillos and the substitutability of flavored versus unflavored disposable e-cigarettes between young adult sexual and gender minorities (SGM) and heterosexual females. SGM female cigarillousers will be recruited from participants of the Supplemental Aim 1 sample and be compared to heterosexual female participants of the parent study (or Aim 3). Both samples will receive the same questions and be exposed to the same ETM conditions tocompare perceptions of appeal of flavors and substitutability between cigarillos, e-cigarettes, and other tobacco products.

ELIGIBILITY:
Aim 1:

Inclusion Criteria:

* Age range: 21-28 years
* Individuals who have smoked an average of 2 cigarillos per week over the past month.
* Individuals willing to provide informed consent and participate in the online survey.

Exclusion Criteria:

- Individuals who have never smoked a cigarillo

Supplemental Aim 1:

Inclusion Criteria:

* Age range: 21-28 years
* Individuals who have smoked an average of 2 cigarillos per week over the past month.
* Individuals willing to provide informed consent and participate in the online survey.
* Individuals who identify as female, trans-female/woman, or non-binary
* Individuals who identify as not heterosexual

Exclusion Criteria:

* Individuals who currently do not smoke at least 2 cigarillos per week
* Individuals who identify as male or trans-man
* Individuals who identify as heterosexual

Supplemental Aim 1 Interviews:

Inclusion Criteria

* Previous participant in Supplemental Aim 1 or Aim 1 survey.
* Participant agreed to be contacted to participate in future studies.
* Individuals who have ever used a cigarillo.
* Individuals willing to provide informed consent and participate in the interview.
* Individuals who identify as women (cis- or transwomen)

Exclusion Criteria:

* Individuals who have never used a cigarillo.
* Individuals who do not identify as women (cis- or transwomen)
* Individuals unwilling to provide informed consent and participate in the interview

Cognitive Interviews:

Inclusion Criteria:

* Age range: 21-28 years
* Sample 1: Individuals who have smoked an average of 2 cigarillos per week over the past month and did not smoke an average of 2 e-cigarettes per week over the past month
* Sample 2: Individuals who have smoked an average of 2 e-cigarettes per week over the past month and did not smoke an average of 2 cigarillos per week over the past month
* Sample 3: Individuals who have smoked an average of 2 cigarillos AND 2 e-cigarettes per week over the past month
* Sample 4: Individuals who have never smoked tobacco or used nicotine products
* Individuals willing to provide informed consent and participate in a qualitative interview.

Aim 2:

Inclusion Criteria

* Age range: 16-28 years
* Individuals not having chronic eye diseases known to interfere with eye tracking equipment (i.e. glaucoma, regression lenses, cataracts, etc.)
* Individuals willing to meet in-person at lab in Columbus, Ohio to complete study procedures.
* Individuals willing to provide informed consent or assent and participate in the online survey.

Exclusion Criteria:

- Pregnant females

Aim 3:

Inclusion Criteria:

* Age range: 21-28 years
* Individuals who smoked 2 cigarillos per week over the past month.

Exclusion Criteria:

* Individuals who currently do not smoke at least 2 cigarillos per week
* Females who are pregnant or lactating

Supplemental Aim 3:

Inclusion Criteria:

* Age range: 21-28 years
* Individuals who smoked 2 cigarillos a week over the past month
* Individuals who identify as female, trans-female/woman, or non-binary
* Individuals who identify as lesbian, bisexual, pansexual, or queer

Exclusion Criteria:

* Individuals who currently do not smoke at least 2 cigarillos per week
* Individuals who identify as male or transman
* Individuals who identify as heterosexual

Ages: 16 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 658 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Appeal scores of flavored versus unflavored cigarillos in cigarillo users based on initial online survey scores | At baseline
  Within-subjects analyses (one sample paired t-tests) will be used to assess appeal scores of flavored versus unflavored cigarillos in cigarillo users based on initial online survey scores.
  Appeal Scores are on a 7-point LIKERT Scale from Strongly Disagree to Strongly Agree for three indicators. High values indicate higher greater appeal while low values indicate lower appeal.
Appeal scores of flavored cigarillos versus flavored e-cigarettes in cigarillo users based on initial online survey scores | At baseline
  Within-subjects analyses (one sample paired t-tests) will be used to assess appeal scores of flavored cigarillos versus flavored e-cigarettes in cigarillo users based on initial online survey scores.
  Appeal Scores are on a 7-point LIKERT Scale from Strongly Disagree to Strongly Agree for three indicators. High values indicate higher greater appeal while low values indicate lower appeal.
Perceptions of harm of flavored cigarillos versus unflavored cigarillos in cigarillo users as assessed by initial online survey scores | At baseline
  Within-subjects analyses (one sample paired t-tests) will be used to assess perceptions of harm of flavored cigarillos versus unflavored cigarillos in cigarillo users as assessed by initial online survey scores.
  Perception of Harm scores are on a 3-point scale: Less harmful, about the same level (or as harmful), and more harmful. Higher values indicate more perceived harm while lower values indicate less perceived harm.
Visual attention as assessed by dwell time visual attention on product packages | Immediately after exposure to product advertisements
  Visual attention as assessed by dwell time visual attention on product packages across a set of only flavored, only unflavored or mixed flavor advertisements
Attentional bias in flavored cigarillos products versus unflavored cigarillo advertisements | Immediately after exposure to product advertisements
  Attentional bias in flavored cigarillos products versus unflavored cigarillo advertisements. Attentional bias is defined as greater duration of attention to flavored stimuli.
Abuse liability of flavored cigarillos products versus unflavored cigarillo as measured by Sensitivity (alpha) | One week after exposure to product advertisements
  Abuse liability of flavored cigarillos products versus unflavored cigarillo as measured by sensitivity (alpha): The sensitivity of demand and the measure of cigarillo purchasing across the price function.
Abuse liability of flavored cigarillos products versus unflavored cigarillo as measured by intensity (Q0) | One week after exposure to product advertisements
  Abuse liability of flavored cigarillos products versus unflavored cigarillo as measured by Intensity (Q0): The intensity of demand and level of cigarillo purchasing at the lowest cost
Substitutability of flavored e-cigarettes versus unflavored e-cigarettes | One week after exposure to product advertisements
  Substitutability of flavored e-cigarettes versus unflavored e-cigarettes. To analyze the level of substitution of alternative tobacco products, the study team will fit linear regressions for each product type. Consistent with previous research slopes that significantly differ from zero will be considered substitutes.
Degree of substitutability of flavored e-cigarettes when compared to various cigarillo flavors | One week after exposure to product advertisements
  Degree of substitutability of flavored e-cigarettes when compared to various cigarillo flavors.
  To analyze the level of substitution of alternative tobacco products, the study team will fit linear regressions for each product type. Consistent with previous research slopes that significantly differ from zero will be considered substitutes. To compare substitutability in the four flavors, slopes will be compared across the four ETM conditions using one-way ANOVA
Future use intentions of flavored cigarillos products versus unflavored cigarillo advertisements | One week after exposure to product advertisements
  Future use intentions of flavored cigarillos products versus unflavored cigarillo advertisements.
  Future Use Intentions are scored on a 4-point scale: Definitely not, probably not, probably yes, definitely yes. Higher values indicate greater intention to use tobacco product(s) and lower values indicate lower intention to use tobacco product(s)
Perceptions of harm of flavored cigarillos products versus unflavored cigarillo advertisements | Immediately after exposure to product advertisements
  Perceptions of harm of flavored cigarillos products versus unflavored cigarillo advertisements (assessed on absolute and relative risk scales).
  Perception of Harm scores are on a 3-point scale: Less harmful, about the same level (or as harmful), and more harmful. Higher values indicate more perceived harm while lower values indicate less perceived harm.
Perceptions of harm of flavored cigarillos products versus unflavored cigarillo advertisements | One week after exposure to product advertisements
  Perceptions of harm of flavored cigarillos products versus unflavored cigarillo advertisements (assessed on absolute and relative risk scales).
  Perception of Harm scores are on a 3-point scale: Less harmful, about the same level (or as harmful), and more harmful. Higher values indicate more perceived harm while lower values indicate less perceived harm.
Product use intentions at the one- week follow-up survey | One week after exposure to product advertisements
  Product use intentions (any/none) at the one- week follow-up survey
Appeal ratings of flavored cigarillos products versus unflavored cigarillo advertisements | One week after exposure to product advertisements
  Appeal ratings of flavored cigarillos products versus unflavored cigarillo advertisements.
  Appeal Scores are on a 7-point LIKERT Scale from Strongly Disagree to Strongly Agree for three indicators. High values indicate higher greater appeal while low values indicate lower appeal.
Minnesota Tobacco Withdrawal Scale | At baseline and immediately after ETM
  Participants evaluate themselves on eight DSM-5 symptoms associated with tobacco withdrawal on a five-point scale from None to Severe and each item is scored from 0 (None) to 4 (Severe). Total scores range from 0 to 32 on this scale with higher scores indicating greater levels of withdrawal.
Nicotine Dependence - Aim 1 survey | At baseline
  Participants report their level of agreement with twelve statements related to nicotine dependence on a five-point Likert scale from Never to Always. Total scores range from 0 to 60 with higher scores indicating greater nicotine dependence.
  Also asked on Aim 1 Survey
Nicotine Dependence - Aim 3/Supplemental Aim 3 group | At baseline and immediately after ETM
  Participants report their level of agreement with twelve statements related to nicotine dependence on a five-point Likert scale from Never to Always. Total scores range from 0 to 60 with higher scores indicating greater nicotine dependence.
  Also asked on Aim 1 Survey
Likelihood of flavor use - Aim 1 survey | At baseline
  Participants are asked how likely they are to use six flavors of cigarillos on a four-point scale from Definitely Never Use to Regularly Use.
Likelihood of flavor use - Aim 3/Supplemental Aim 3 group | At baseline and immediately after ETM
  Participants are asked how likely they are to use six flavors of cigarillos on a four-point scale from Definitely Never Use to Regularly Use.
Perceptions of flavors - Aim 1 survey | At baseline
  Participants are asked their perceptions of six different cigarillo flavors on a six-point scale from Very Bad (1) to Very Good (6). Also asked on Aim 1 Survey.
  Each item will receive a rating from 1 (Very Bad) to 6 (Very Good), but these will not be added together in a scale
Perceptions of flavors - Aim 3/Supplemental Aim 3 group | At baseline and immediately after ETM
  Participants are asked their perceptions of six different cigarillo flavors on a six-point scale from Very Bad (1) to Very Good (6). Also asked on Aim 1 Survey.
  Each item will receive a rating from 1 (Very Bad) to 6 (Very Good), but these will not be added together in a scale

CONTACTS AND LOCATIONS:
Overall Officials: Erika Trapl, PhD, Principal Investigator — Case Western Reserve University, Case Comprehensive Cancer Center
Locations (1):
- Case Western Reserve University, Case Comprehensive Cancer Center, Cleveland, Ohio, United States